CLINICAL TRIAL: NCT02756494
Title: Some Biomarkers Underlying in Ischemic Stroke in Chinese Young Adults: a Protocol for a Case-control Clinical Trial
Brief Title: Ischemic Stroke in Chinese Young Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Director, Head of Endocrinology, Principal Investigator, Beijing Chao Yang Hospital
Other Study IDs: Ischemic201603
Record Dates: First submitted 2016-04-03; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ischemic Stroke in Young Adults: Patients between 18 and 45 years of age with a first ever ischaemic stroke are eligible for this study from the Department of Beijing Chaoyang Hospital between January 1, 2016 and December 31, 2016. All patients were defined as a sudden loss of global or focal cerebral function that persisted with a probable vascular cause for 24h and confirmed by brain CT or MRI.
  Interventions: Biological: Ischemic Stroke
- matched control subjects: The age-, sex-, and time of enrollment-matched control cohort was randomly identified after eliminating the study subjects and those who had been given a diagnosis of any stroke at any time.
  Interventions: Biological: Ischemic Stroke

INTERVENTIONS:
Biological: Ischemic Stroke — Ischemic Stroke in Chinese Young Adults

SUMMARY:
Stroke is the fifth leading cause of death in the United States and the leading cause of disability. However, in China, stroke is one of the most frequent causes of death and chronic disability. Ischemic strokes in adults younger than 45 years of age were regarded as a relatively uncommon event in the proportion of <5% of all ischemic strokes.

DETAILED DESCRIPTION:
Currently, stroke is the fifth leading cause of death in the United States and the leading cause of disability. However, in China, stroke is one of the most frequent causes of death and chronic disability. Ischemic strokes in adults younger than 45 years of age were regarded as a relatively uncommon event in the proportion of <5% of all ischemic strokes. Our study aimed to evaluate some Biomarkers Underlying in Ischemic Stroke in Chinese Young Adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 45 years of age with a first ever ischaemic stroke are eligible for this study from the Department of Beijing Chaoyang Hospital between January 1, 2016 and December 31, 2016.
* All patients were defined as a sudden loss of global or focal cerebral function that persisted with a probable vascular cause for 24h and confirmed by brain CT or MRI.

Exclusion Criteria:

* The exclusion criteria will include patients with intracranial lesions or cerebrovascular disease (including cerebral venous sinus thrombosis)
* History that have caused sequelae, such as movement disorders, mood disorders, cognitive dysfunction or speech problems; or individuals who are pregnant or breast feeding.
* Patients with serious diseases that are related to the heart, liver, kidney or haematopoietic system will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between 18 and 45 years of age with a first ever ischaemic stroke are eligible for this study from the Department of Beijing Chaoyang Hospital between January 1, 2016 and December 31, 2016. All patients were defined as a sudden loss of global or focal cerebral function that persisted with a probable vascular cause for 24h and confirmed by brain CT or MRI.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of Ischemic Stroke in Chinese Young Adults | every two months, up to 24 months
  the incidence of Ischemic Stroke

IPD SHARING:
Plan to Share IPD: Undecided